CLINICAL TRIAL: NCT03884803
Title: Healthy Moms for Healthy Babies: Implementation of an Enhanced E-Health Prenatal Program to Promote Maternal Mental Health
Brief Title: Healthy Moms for Healthy Babies
Acronym: HealthyMoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University (Other)
Collaborators: Medtech-Fonds de soutien à l'innovation en santé et en services sociaux (FSISSS) (Unknown)
Responsible Party: Principal Investigator, Deborah Da Costa, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MP-37-2019-5119
Record Dates: First submitted 2019-03-15; First posted 2019-03-21 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HealthyMoms web-based program (Other): An on-line self-help psychoeducational website for new moms that includes educational learning modules and tools to prevent/reduce depression. .
  Interventions: Behavioral: E-health website
- Control group (Other): No access to the intervention but to continue with standard care. Will complete the same questionnaires as the HealthyMoms group.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: E-health website — Access to the e-health intervention (website)
  Arms: HealthyMoms web-based program
Other: Standard Care — Control group to continue with standard care
  Arms: Control group

SUMMARY:
HealthyMoms is prototype website with accurate and easily accessible information on the impact of depression, anxiety and stress during pregnancy and the importance of healthy behaviours (physical activity, nutrition, sleep). This clinical trial is to pilot test the implementation of the e-health intervention alongside standard antenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate in French or English
* At least 18 years of age
* First child
* Internet and email access

Exclusion Criteria:

* Do not meet inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Acceptability of healthymoms website | 6 weeks post intervention
  Determine the acceptability of the program in terms of uptake, adherence, and user satisfaction. To use the Satisfaction and Usability survey
Change from baseline on depressed mood | study entry, 6 weeks post intervention, 3 months post delivery, 6 months post delivery
  Estimate the range of effect sizes for depressive symptoms in order to evaluate the efficacy of the program (healthymoms website). Measured by the Edinburgh Postnatal Depression Scale.

SECONDARY OUTCOMES:
Changes from baseline on pregnancy related anxiety | study entry, 6 weeks post intervention
  Evaluate changes in pregnancy related anxiety in order to evaluate the efficacy of the healthymoms website. Using the Pregnancy-related Anxiety questionnaire-revised (PRAQ-R)
Changes from baseline in physical activity | study entry, 6 weeks post intervention, 3 months post delivery, 6 months post delivery
  Evaluate changes in a health behaviour (physical activity) in order to evaluate the efficacy of the healthymoms website. Use of the International Physical Activity Questionnaire-Short Form (IPAQ-SF)
Changes from baseline on sleep quality | study entry, 6 weeks post intervention, 3 months post delivery, 6 months post delivery
  Evaluate changes in a health behaviour (sleep quality) in order to evaluate the efficacy of the healthymoms website. Use of the Pittsburgh Sleep Quality Index-short
Changes from baseline regarding satisfaction with antenatal care | study entry, 6 weeks post intervention
  Evaluate the changes in satisfaction with antenatal care in order to inform future implementation of the healthymoms website

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada